CLINICAL TRIAL: NCT04569409
Title: Phase 3 Clinical Study to Evaluate Efficacy and Safety of ALLO-ASC-DFU in Patients With Diabetic Wagner Grade 2 Foot Ulcers: A Randomized, Comparator-controlled, Double-blind, Parallel-group, Multi-center Study
Brief Title: Clinical Study to Evaluate Efficacy and Safety of ALLO-ASC-DFU in Patients With Diabetic Wagner Grade 2 Foot Ulcers.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLO-ASC-DFU-302
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-12

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ALLO-ASC-DFU (Experimental): Hydrogel sheet containing allogenic adipose-derived mesenchymal stem cells
  Interventions: Biological: ALLO-ASC-DFU
- Vehicle sheet (Placebo Comparator): Hydrogel sheet without allogenic mesenchymal stem cell
  Interventions: Procedure: Vehicle Sheet

INTERVENTIONS:
Biological: ALLO-ASC-DFU — Application of ALLO-ASC-DFU sheet to Diabetic Wagner grade 2 Foot Ulcer
  Arms: ALLO-ASC-DFU
Procedure: Vehicle Sheet — Application of Vehicle sheet to Diabetic Wagner grade 2 Foot Ulcer
  Arms: Vehicle sheet

SUMMARY:
This is a phase III double-blind study to evaluate the efficacy and safety of ALLO-ASC-DFU in patients with Diabetic Wagner grade 2 Foot Ulcer, compared to placebo therapy.

DETAILED DESCRIPTION:
Experimental: ALLO-ASC-DFU, Placebo Comparator: Vehicle Sheet, Study type: Interventional, Study design: Randomized, Placebo-controlled, Double blind, Parallel-group, Multi-center Study

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between 19 and 75 years of age.
2. Subject is diagnosed with Type I or Type II diabetics.
3. Diabetic foot ulcer has been more than 4 weeks but less than 52 weeks at the screening visit.
4. Ulcer located in the foot and ulcer size is between 1.5~15 cm2.
5. Ulcer graded 2 by Wagner grade.
6. Foot ulcer extended to ligament, tendon, joint capsule, fascia, muscle and periosteum.
7. Ulcer is free of necrotic debris.
8. Ulcer area blood circulation meets one of the following criteria;

   * Blood vessels around the ulcer detected by Doppler Test
   * Range of Ankle Brachial Index (ABI) is > 0.7 to < 1.3
   * Transcutaneous Oxygen Pressure (TcPO2) > 30mmHg or Toe Blood Pressure (TBP) > 40mmHg.
   * Skin Perfusion Pressure (SPP) > 30mmHg
9. Subject is able to give written informed consent prior to study start and willing to comply with the study requirements.

Exclusion Criteria:

1. Ulcer is of non-diabetic pathophysiology.
2. There is gangrene in any part of the target foot ulcer.
3. The longest dimension of the target foot ulcer exceeds 15 cm at the enrollment visit.
4. Other wounds within 2cm of the target foot ulcer.
5. The ulcer has increased or decreased in size by ≥ 30% during two weeks after the screening visit.
6. Patient requiring intravenous (IV) antibiotics to treat foot wound infection at the screening and enrollment visit.
7. Current evidence of active charcot on the study foot, osteomyelitis, cellulitis, or evidence of other infection including fever or purulent drainage from wound site.
8. Patient with skin lesion confirmed by biopsy (when Investigator deems suspicious) and then judged by Investigator to be an etiology other than diabetic foot ulcer.
9. An active malignant tumor(malignant melanoma, squamous cell carcinoma, basal cell carcinoma) on the body or skin.
10. Have a glycated hemoglobin A1c (HbA1c) level of > 14%
11. Have random blood sugar > 450mg/dL
12. Have severe renal failure with creatinine > 3.0mg/dL.
13. Have severe hepatic deficiencies

    * Total bilirubin ≥ 1.5×upper normal limit(UNL)
    * AST, ALT ≥ 2.0×UNL
    * Serum albumin < 2.0mg/dL
14. Is Human Immunodeficiency Virus (HIV) positive
15. Have a known history of allergic or hypersensitive reaction to bovine-derived proteins or fibrin glue
16. Pregnant or breast-feeding.
17. Is unwilling to use an acceptable method of birth control during the whole study.
18. Have a clinically relevant history of alcohol or drugs abuse at the screening visit.
19. Is not able to understand the objective of the study or to comply with the study requirements
20. Is considered by the Investigator to have a significant disease which might impact the study
21. Is considered not suitable for the study by Investigator
22. Have a history of malignancy within the last 5 years (except carcinoma in situ)
23. Is currently or were enrolled in another clinical study within 60 days of screening
24. Have undergone wound treatments with growth factors, dermal substitutes, or other biological therapies within the last 30 days.
25. Is receiving oral or parenteral corticosteroids, any immunosuppressive, or cytotoxic agents with unstable dose within the last 30 days
26. Cannot maintain off-loading process and device.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Proportions of subjects who achieved complete wound closure | During 12 weeks

SECONDARY OUTCOMES:
Time taken to complete wound closure | During 12 weeks
Proportions of subjects who achieved complete wound closure at every visit | During 12 weeks
Change rates in wound size and depth compared to baseline groups | During 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: SeungKyu Han, MD. Ph D, Principal Investigator — Korea University Guro Hospital; BaekKyu Kim, MD. Ph D, Principal Investigator — Seoul National University Bundang Hospital; JunPio Hong, MD. Ph D, Principal Investigator — Asan Medical Center; JiUng Bak, MD. Ph D, Principal Investigator — Borame Medical Center; YeongCheol Seo, MD. Ph D, Principal Investigator — Bucheon St. Mary's Hospital
Locations (5):
- South Korea (5):
  - Bucheon ST. Mary's Hospital, Gyeonggi-do, Bucheon
  - Seoul National University Bundang Hospital, Gyeonggi-do, Seongnam-si
  - Asan Medical Center, Seoul, Seoul
  - Borame Medical Center, Seoul, Seoul
  - Korea University Guro Hospital, Seoul, Seoul

IPD SHARING:
Plan to Share IPD: Undecided